CLINICAL TRIAL: NCT07345962
Title: Assessment of the Expectations and Fears of Pregnant Patients Monitored at the CMCO Regarding Ambulatory Epidural Anesthesia
Acronym: Déambu-Péri
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9946
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ambulatory Epidural
Keywords: Ambulatory epidural; Epidural Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ambulatory epidural anesthesia is a technique that has been described since the late 1990s and has been rapidly gaining popularity in recent years.

Although there is currently no change in the obstetric process, this technique has been shown to improve maternal satisfaction.

Ambulatory epidural s are not yet offered in the maternity wards of Strasbourg University Hospitals.

However, a protocol is currently being studied and should be rolled out soon at the maternity ward of the Centre Médico-chirurgical Obstétrique (CMCO).

This study aims to assess the general interest in this technique among the population concerned.

It also seeks to highlight any fears patients may have that could hinder the implementation of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥18 years old)
* Pregnant women monitored at the CMCO

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult pregnant women monitored at the CMCO
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who expressed interest in ambulatory epidural anesthesia | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation médecine Péri-Opératoire - CHU de Strasbourg - France, Strasbourg, France